CLINICAL TRIAL: NCT00747396
Title: The Bucharest Early Intervention Project: Effects of Early Psychosocial Deprivation on Mental Health in Adolescence
Brief Title: The Bucharest Early Intervention Project
Acronym: BEIP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charles Alexander Nelson III (Other)
Collaborators: Tulane University Health Sciences Center (Other); University of Maryland (Other); University of Minnesota (Other); Temple University (Other); Duke University (Other); MacArthur Foundation (Other); National Institute of Mental Health (NIMH) (NIH); Vanderbilt University (Other); Harvard University (Other); University of North Carolina, Chapel Hill (Other); University of Toronto (Other)
Responsible Party: Sponsor-Investigator, Charles Alexander Nelson III, Richard David Scott Chair in Pediatric Developmental Medicine Research, Professor of Pediatrics and Neuroscience, Boston Children's Hospital
Organization: Boston Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB-P00011741; R01MH091363 (NIH)
Record Dates: First submitted 2008-09-04; First posted 2008-09-05 (Estimated); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Cognitive Ability, General; Psychiatric and/or Mood Disorders; Brain Function; Social Cognition; Health Behavior; Risk-Taking; Executive Function
Keywords: Romania,; children,; foster care,; institutionalization,; brain function,; MRI,; attachment,; language,; growth,; Intelligence Quotient (IQ),; psychiatric symptomatology; early intervention
MeSH Terms: conditions — Health Behavior; Risk-Taking; Language

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Foster Care Placement Group (Experimental): Children randomized to this group were placed in high quality foster care developed for the study.
  Interventions: Other: Foster Care Placement
- Care As Usual Group (No Intervention): Children randomized to this group remained in institutional care.

INTERVENTIONS:
Other: Foster Care Placement — A group of children living in institutions in Bucharest, Romania was randomly assigned to placement in foster care. Foster parents were recruited, consented to background checks, and trained in Romanian. Before placement, foster parents visited their children to begin developing a relationship with the child. Hired foster parents were supported and monitored by project social workers. Foster parents in the BEIP network received frequent visits from the social workers, with visits occurring weekly for several months after placement of the child, then biweekly and later monthly. Foster parents were invited to participate in a support group organized by social workers. Project social workers consulted weekly with US staff experienced in dealing with young children in foster care.
  Other Names: Foster Care Group
  Arms: Foster Care Placement Group

SUMMARY:
The purpose of this study is to determine the long term effects of early intervention (placement into foster care) on physical, cognitive, social and brain development and psychiatric symptomatology in previously institutionalized children.

DETAILED DESCRIPTION:
The Bucharest Early Intervention Project (BEIP) was a randomized controlled trial of foster care as an intervention for children abandoned at or around the time of birth and placed in one of six institutions for young children in Bucharest, Romania (Zeanah et al., 2003). The PI (Nelson) and Co-PIs (Zeanah and Fox) conducted this study beginning in the fall of 2000 from baseline assessments and implementation of the intervention in the spring of 2001.

The BEIP began with comprehensive assessments of 136 institutionalized children and their caregiving environments prior to randomization. Half the children were randomly assigned to high-quality foster care and the other half to remain in institutional care. The average age at foster care placement was 22 months (range=6-31 months). All children were initially seen prior to randomization and again for follow-up assessments at 30 months, 42 months 54 months, 8 years, 12 year and 16 years of age. The development of children in foster care was compared to the development of children in institutions and to a group of never institutionalized children (community controls). These children, now young adults are being assessed at age 21 years.

ELIGIBILITY:
Inclusion Criteria for assessment at age 21 years:

* previously institutionalized and community children that took part in previous BEIP assessments
* target recruitment age is +/- 6 mos of 21st birthday

Exclusion Criteria for assessment at age 21 years:

* open or closed head injury within the past 12 months
* viral or bacterial meningitis within the past 12 months

Ages: 21 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 136 (Actual)
Dates: Start 2000-09 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Changes in EEG Coherence Brain Function | baseline, 30 mos, 42 mos, 8 years, 12 years, 16 years, 21 years
  EEG coherence
Changes in EEG Power Brain Function | baseline, 30 mos, 42 mos, 8 years, 12 years, 16 years, 21 years
  EEG power
Changes in EEG Asymmetry Brain Function | baseline, 30 mos, 42 mos, 8 years, 12 years, 16 years, 21 years
  EEG asymmetry
Changes in Attachment Disturbances and Disorders | baseline, 30 mos, 42 mos, 54 mos, 8 years, 12 years, 16 years
  Disturbances of Attachment Interview
Changes in Attachment Style | baseline, 30 mos and 42 mos
  Strange Situation Procedure
Changes in Cognition in later childhood and adolescence | 8 years, 12 years, 16-18 years
  Wechsler Intelligence Scale for Children-IV
Changes in Cognition in young adulthood | 21 years
  Wechsler Adult Intelligence Scale
Changes in Cognition in early childhood | baseline, 30 months, 42 months
  Bayley Scales of Infant Development
Changes in weight | baseline, 30 mos, 42 mos, 8 years, 12 years, 16 years, 21 years
  weight in kilograms
Changes in height | baseline, 30 mos, 42 mos, 8 years, 12 years, 16 years, 21 years
  Height measured in centimeters
Changes in head circumference | baseline, 30 mos, 42 mos, 8 years, 12 years, 16 years, 21 years
  Head circumference in centimeters
Changes in Psychiatric Symptomatology in adolescence | 12 years, 16 years
  Diagnostic Interview Schedule for Children -IV
Changes in Psychiatric Symptomatogology | 54 months, 8 years
  Preschool And Child Adolescent Psychological Assessment
Changes in Psychiatric Symptomatogology | 21 years
  Diagnostic Interview Schedule + Substance Abuse Module
Changes in Expressive Language Quality | 30 mos, 42 mos and 8 years
  language sample from interview
Changes in Caregiving Environment | baseline, 30 mos and 42 mos
  Observational Record of Caregiving Environment
Changes in Indiscriminate Behavior | 54 mos, 8 years and 12 years
  Stranger at the Door
Changes in Emotion Discrimination | baseline, 30 mos, 42 mos and 8 years
  Event-related Potentials
Changes in Face Recognition | baseline, 30 mos, 42 mos and 8 years
  Event-related Potentials
Changes in Brain Structure | 8 years, 16 years, 21 years
  MRI
Changes in Problem Behaviors | baseline, 30 mos and 42 mos
  Infant Toddler Social Emotional Assessment
Changes in Social Communication and Interaction | baseline, 30 mos, 42 mos, 8 years, 12 years, 16 years
  Social Communication Questionnaire
Changes in Genetics | 8 years, 12 years, 16 years
  Buccal Swab

SECONDARY OUTCOMES:
Changes in Emotional Reactivity/Temperament | baseline, 30 mos and 42 mos
  Laboratory Temperament Assessment Battery (Lab-TAB) Puppets and Peek-a-boo
Motor Skills | 8 years
  Bruininks-Oseretsky Test-2

OTHER OUTCOMES:
Changes in Physiological Reactivity to Stress | 12 years, 16 years
  Trier Social Stress Test

CONTACTS AND LOCATIONS:
Overall Officials: Charles A Nelson, Ph.D., Principal Investigator — Children's Hospital Boston/Harvard University; Nathan A. Fox, Ph.D., Principal Investigator — University of Maryland; Charles H. Zeanah, M.D., Principal Investigator — Tulane University Health Sciences Center
Locations (1):
- Fundatia Tanner, Bucharest, Romania

REFERENCES:
- [Derived] Arnett AB, Antunez M, Zeanah C, Fox NA, Nelson CA. Physical and neurophysiological maturation associated with ADHD among previously institutionalized children: a randomized controlled trial. J Child Psychol Psychiatry. 2025 Jul;66(7):967-979. doi: 10.1111/jcpp.14110. Epub 2025 Jan 11. PMID 39797613
- [Derived] Guyon-Harris KL, Plamondon A, Humphreys KL, Wade M, Gleason MM, Tibu F, Nelson CA, Fox NA, Zeanah CH. Structure of Psychopathology in Romanian Preschool-Aged Children in an Epidemiological and a High-Risk Sample. JAACAP Open. 2023 Nov;1(3):173-183. doi: 10.1016/j.jaacop.2023.06.004. Epub 2023 Jul 19. PMID 38500494
- [Derived] King LS, Guyon-Harris KL, Valadez EA, Radulescu A, Fox NA, Nelson CA, Zeanah CH, Humphreys KL. A Comprehensive Multilevel Analysis of the Bucharest Early Intervention Project: Causal Effects on Recovery From Early Severe Deprivation. Am J Psychiatry. 2023 Aug 1;180(8):573-583. doi: 10.1176/appi.ajp.20220672. Epub 2023 May 22. PMID 37211832
- [Derived] Humphreys KL, Guyon-Harris KL, Tibu F, Wade M, Nelson CA, Fox NA, Zeanah CH. Psychiatric outcomes following severe deprivation in early childhood: Follow-up of a randomized controlled trial at age 16. J Consult Clin Psychol. 2020 Dec;88(12):1079-1090. doi: 10.1037/ccp0000613. PMID 33370132
- [Derived] Humphreys KL, Machlin LS, Guyon-Harris KL, Nelson CA, Fox NA, Zeanah CH. Psychosocial deprivation and receptive language ability: a two-sample study. J Neurodev Disord. 2020 Dec 16;12(1):36. doi: 10.1186/s11689-020-09341-2. PMID 33327936
- [Derived] Slopen N, Tang A, Nelson CA, Zeanah CH, McDade TW, McLaughlin KA, Fox NA. The Consequences of Foster Care Versus Institutional Care in Early Childhood on Adolescent Cardiometabolic and Immune Markers: Results From a Randomized Controlled Trial. Psychosom Med. 2019 Jun;81(5):449-457. doi: 10.1097/PSY.0000000000000696. PMID 31008902
- [Derived] Wade M, Fox NA, Zeanah CH, Nelson CA, Drury SS. Telomere Length and Psychopathology: Specificity and Direction of Effects Within the Bucharest Early Intervention Project. J Am Acad Child Adolesc Psychiatry. 2020 Jan;59(1):140-148.e3. doi: 10.1016/j.jaac.2019.02.013. Epub 2019 Mar 4. PMID 30844465
- [Derived] Wade M, Fox NA, Zeanah CH, Nelson CA. Effect of Foster Care Intervention on Trajectories of General and Specific Psychopathology Among Children With Histories of Institutional Rearing: A Randomized Clinical Trial. JAMA Psychiatry. 2018 Nov 1;75(11):1137-1145. doi: 10.1001/jamapsychiatry.2018.2556. PMID 30267045
- [Derived] Johnson DE, Tang A, Almas AN, Degnan KA, McLaughlin KA, Nelson CA, Fox NA, Zeanah CH, Drury SS. Caregiving Disruptions Affect Growth and Pubertal Development in Early Adolescence in Institutionalized and Fostered Romanian Children: A Randomized Clinical Trial. J Pediatr. 2018 Dec;203:345-353.e3. doi: 10.1016/j.jpeds.2018.07.027. Epub 2018 Aug 29. PMID 30172435
- [Derived] Humphreys KL, Miron D, McLaughlin KA, Sheridan MA, Nelson CA, Fox NA, Zeanah CH. Foster care promotes adaptive functioning in early adolescence among children who experienced severe, early deprivation. J Child Psychol Psychiatry. 2018 Jul;59(7):811-821. doi: 10.1111/jcpp.12865. Epub 2018 Feb 1. PMID 29389015
- [Derived] Humphreys KL, McGoron L, Sheridan MA, McLaughlin KA, Fox NA, Nelson CA 3rd, Zeanah CH. High-Quality Foster Care Mitigates Callous-Unemotional Traits Following Early Deprivation in Boys: A Randomized Controlled Trial. J Am Acad Child Adolesc Psychiatry. 2015 Dec;54(12):977-83. doi: 10.1016/j.jaac.2015.09.010. Epub 2015 Oct 9. PMID 26598472
- [Derived] Humphreys KL, Gleason MM, Drury SS, Miron D, Nelson CA 3rd, Fox NA, Zeanah CH. Effects of institutional rearing and foster care on psychopathology at age 12 years in Romania: follow-up of an open, randomised controlled trial. Lancet Psychiatry. 2015 Jul;2(7):625-34. doi: 10.1016/S2215-0366(15)00095-4. Epub 2015 Jun 23. PMID 26303560
- [Derived] Bick J, Zhu T, Stamoulis C, Fox NA, Zeanah C, Nelson CA. Effect of early institutionalization and foster care on long-term white matter development: a randomized clinical trial. JAMA Pediatr. 2015 Mar;169(3):211-9. doi: 10.1001/jamapediatrics.2014.3212. PMID 25622303
- [Derived] Gleason MM, Fox NA, Drury S, Smyke A, Egger HL, Nelson CA 3rd, Gregas MC, Zeanah CH. Validity of evidence-derived criteria for reactive attachment disorder: indiscriminately social/disinhibited and emotionally withdrawn/inhibited types. J Am Acad Child Adolesc Psychiatry. 2011 Mar;50(3):216-231.e3. doi: 10.1016/j.jaac.2010.12.012. Epub 2011 Feb 1. PMID 21334562
- [Derived] Bos KJ, Zeanah CH Jr, Smyke AT, Fox NA, Nelson CA 3rd. Stereotypies in children with a history of early institutional care. Arch Pediatr Adolesc Med. 2010 May;164(5):406-11. doi: 10.1001/archpediatrics.2010.47. PMID 20439790
- [Derived] Johnson DE, Guthrie D, Smyke AT, Koga SF, Fox NA, Zeanah CH, Nelson CA 3rd. Growth and associations between auxology, caregiving environment, and cognition in socially deprived Romanian children randomized to foster vs ongoing institutional care. Arch Pediatr Adolesc Med. 2010 Jun;164(6):507-16. doi: 10.1001/archpediatrics.2010.56. Epub 2010 Apr 5. PMID 20368481